CLINICAL TRIAL: NCT03310580
Title: A Prospective, Double-masked, Randomized, Multicenter, Placebo-controlled, Parallel-group Study Assessing the Safety and Ocular Hypotensive Efficacy and Optimum Concentration to be Used Clinically of Netarsudil Ophthalmic Solution in Japanese/Japanese-American Subjects With Open-angle Glaucoma or Ocular Hypertension in the United States
Brief Title: Study of Netarsudil Ophthalmic Solution in Japanese/Japanese-American Subjects With Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR-13324-CS205
Record Dates: First submitted 2017-10-13; First posted 2017-10-16 (Actual); Results first posted 2019-11-15 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Primary Open Angle Glaucoma or Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AR-13324 Ophthalmic Solution 0.02% (Experimental): Topical sterile ophthalmic solution; 1 drop daily to each eye for 28 days
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.02%
- AR-13324 Ophthalmic Solution 0.04% (Experimental): Topical sterile ophthalmic solution; 1 drop daily to each eye for 28 days
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.04%
- Placebo Comparator (Placebo Comparator): Topical sterile ophthalmic solution; 1 drop daily to each eye for 28 days
  Interventions: Drug: AR-13324 Ophthalmic Solution Placebo

INTERVENTIONS:
Drug: AR-13324 Ophthalmic Solution 0.02% — Administered to each eye, once daily (QD) in the evening (PM) for 28 days
  Arms: AR-13324 Ophthalmic Solution 0.02%
Drug: AR-13324 Ophthalmic Solution 0.04% — Administered to each eye, once daily (QD) in the evening (PM) for 28 days
  Arms: AR-13324 Ophthalmic Solution 0.04%
Drug: AR-13324 Ophthalmic Solution Placebo — Administered to each eye, once daily (QD) in the evening (PM) for 28 days
  Arms: Placebo Comparator

SUMMARY:
To test the safety and effectiveness of AR-13324 0.02% and 0.04% ophthalmic solution relative to placebo in Japanese/Japanese-American subjects with open-angle glaucoma or ocular hypertension in US.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years or older
2. Be of Japanese ethnicity within the 2nd generation defined as (a) 1st generation born in Japan, immigrated to US and (b) 2nd generation - parents are 1st generation and patient was born in US as an American citizen
3. Diagnosis of open-angle glaucoma or ocular hypertension in both eyes
4. Medicated intraocular pressure >/= 15 mmHg and < 30 mmHg in both eyes at screening
5. OAG eyes - unmedicated IOP >/= 15 mmHg and < 35 mmHg at 2 qualification visits at 08:00, 10:00 and 16:00
6. OHT eyes - unmedicated IOP >/= 22 mmHg and < 35mmHg at 08:00, 10:00 and 16:00
7. Best corrected visual acuity + 1.0 logMAR or better by ETDRS in each eye
8. Able to give signed informed consent and follow instructions

Exclusion Criteria:

1. Clinically significant ocular disease
2. Pseudoexfoliation or pigment dispersion component glaucoma, history of angle closure glaucoma or narrow angles
3. Intraocular pressure >/=35 mmHg in either eye
4. Ocular hyperemia score of moderate (+2) at qualification visit #2
5. Previous glaucoma intraocular surgery
6. Refractive surgery in either eye
7. Ocular injury within 6 months prior to screening or ocular surgery or non-refractive laser treatment within 3 months prior to screening
8. Recent or current ocular infection or inflammation in either eye
9. Use of ocular medication in either eye of any kind within 30 days of screening and throughout the study
10. Mean central corneal thickness > 620 µm in either eye
11. Any abnormality preventing reliable applanation tonometry of either eye
12. Known hypersensitivity to benzalkonium chloride or excipients of netarsudil ophthalmic solution
13. Clinically significant abnormalities in screening lab tests
14. Clinically significant systemic disease that might interfere with the study
15. Participated in any investigational study within 30 days prior to screening
16. Systemic medication that could have a substantial effect on IOP within 30 days prior to screening or anticipated during the study
17. Women of child-bearing potential who are pregnant, nursing, planning a pregnancy or not using a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ramirez-Davis, Study Director — Aerie Pharmaceuticals
Locations (40):
- United States (40):
  - Arizona Eye Center, Chandler, Arizona
  - Arizona Glaucoma Specialists, Phoenix, Arizona
  - Milton M. Hom, OD FAAO FACAAISc, Azusa, California
  - Havana Research Institute, Burbank, California
  - Global Research Management, Glendale, California
  - Southern California Eye Physicians & Surgeons, Los Alamitos, California
  - East West Eye Institute, Los Angeles, California
  - USC Roski Eye Institute University of Souther California, Los Angeles, California
  - Global Research Foundation, Los Angeles, California
  - The Eye Research Foundation, Newport Beach, California
  - Southern California Eye Physicians Surgeons, Pasadena, California
  - North Bay Eye Associates Inc., Petaluma, California
  - Martel Eye, Rancho Cordova, California
  - University of California, San Diego, California
  - AdvanceMed Clinical Research, San Diego, California
  - Glaucoma Center of San Francisco, San Francisco, California
  - Samsum Clinic, Santa Barbara, California
  - MCB Clinical Research Centers LLC, Colorado Springs, Colorado
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Jenkins Eye Care, Honolulu, Hawaii
  - Winward Eye Physicians and Eye Surgeons, Kailua, Hawaii
  - Island Eye Care, Inc., Kailua, Hawaii
  - They Eye Care Institute, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Emil A. Stein MD Ltd, Las Vegas, Nevada
  - AdvanceMed Clinical Research, Las Vegas, Nevada
  - New York Eye Infirmary of Mount Sinai, New York, New York
  - The Shimmyo Group, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Optimed Research, Marysville, Ohio
  - Glaucoma Consultants and Center for Eye Research, PA, Mt. Pleasant, South Carolina
  - University Eye Specialists, Maryville, Tennessee
  - VRF Eye Speciality Group, Memphis, Tennessee
  - Lake Travis Eye and Laser Center, Lakeway, Texas
  - DCT - Shah Research LLC dba Discovery Clinical Trials, Mission, Texas
  - Round Rock Eye Consultants, Round Rock, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - R and R Eye Research LLC, San Antonio, Texas
  - Emerson Clinical Research Institute, Falls Church, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- AR-13324 Ophthalmic Solution 0.02%: AR-13324 Ophthalmic Solution 0.02% : Topical sterile ophthalmic solution; 1 drop daily to each eye for 28 days
- AR-13324 Ophthalmic Solution 0.04%: AR-13324 Ophthalmic Solution 0.04%: Topical sterile ophthalmic solution; 1 drop daily to each eye for 28 days
- Placebo Comparator: AR-13324 Ophthalmic Solution Placebo: Topical sterile ophthalmic solution; 1 drop daily to each eye for 28 days
Period: Overall Study
Arm/Group | AR-13324 Ophthalmic Solution 0.02% | AR-13324 Ophthalmic Solution 0.04% | Placebo Comparator
Started | 15 | 15 | 12
Completed | 15 | 14 | 12
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population (ITT)
Groups:
- AR-13324 Ophthalmic Solution 0.02%: AR-13324 Ophthalmic Solution 0.02%: Topical sterile ophthalmic solution; 1 drop daily to each eye for 28 days
- Total: Total of all reporting groups
Arm/Group | AR-13324 Ophthalmic Solution 0.02% | AR-13324 Ophthalmic Solution 0.04% | Placebo Comparator | Total
Number analyzed (Participants) | 14 | 14 | 12 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 6 | 22
  >=65 years | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (20.32) | 60.9 (12.12) | 65.6 (14.98) | 62.4 (15.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 8 | 29
  Male | 4 | 3 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 12 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese 1st Generation | 11 | 12 | 6 | 29
  Japanese 2nd Generation | 3 | 2 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 12 | 40

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal IOP (Intraocular Pressure) (mmHg)
Description: Mean diurnal intraocular pressure (IOP) at week 4, measured by Goldman Applanation Tonometry (GAT).
Time Frame: 28 Days
Population: Intent to treat (ITT) population
Measure: Mean (Standard Error); unit: mmHg
Groups:
- AR-13324 Ophthalmic Solution 0.02%: AR-13324 ophthalmic solution 0.02%; 1 drop daily to each eye for 28 days
  AR-13324 Ophthalmic Solution 0.02%: Topical sterile ophthalmic solution
- AR-13324 Ophthalmic Solution 0.04%: AR-13324 ophthalmic solution 0.04%; 1 drop daily to each eye for 28 days
  AR-13324 Ophthalmic Solution 0.04%: Topical sterile ophthalmic solution
- Placebo Comparator: AR-13324 ophthalmic solution placebo; 1 drop daily to each eye for 28 days
  AR-13324 Ophthalmic Solution Placebo; Topical sterile ophthalmic solution
Arm/Group | AR-13324 Ophthalmic Solution 0.02% | AR-13324 Ophthalmic Solution 0.04% | Placebo Comparator
Number analyzed (Participants) | 14 | 14 | 12
mmHg | 14.35 (0.549) | 14.33 (0.567) | 17.32 (0.576)

2. Secondary Outcome: Extent of Exposure
Description: Exposure to study medication in days for all treatment groups
Time Frame: 28 Days
Population: Exposure to study medication in days for all treatment groups
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AR-13324 Ophthalmic Solution 0.02% | AR-13324 Ophthalmic Solution 0.04% | Placebo Comparator
Number analyzed (Participants) | 15 | 14 | 12
Days | 27.9 (1.91) | 26.8 (7.56) | 27.4 (2.23)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected during the course of the study of 28 days and after 30 days safety follow up
Description: Safety population is defined as all randomized subjects who have received at least 1 dose of study medication.
Arm/Group | AR-13324 Ophthalmic Solution 0.02% | AR-13324 Ophthalmic Solution 0.04% | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 10/15 | 11/14 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AR-13324 Ophthalmic Solution 0.02% (N=15) | AR-13324 Ophthalmic Solution 0.04% (N=14) | Placebo Comparator (N=12)
Conjunctival hyperaemia (Eye disorders) | 10 (10) | 10 (10) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Conjunctival hemorrhage (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Eyelid margin crusting (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Instillation site foreign body sensation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Instillation site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT03310580/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT03310580/SAP_001.pdf